CLINICAL TRIAL: NCT01084538
Title: A One-year, Multicountry, Multicenter Study of Zemplar Injections in Patients With End Stage Chronic Kidney Disease, Undergoing Hemodialysis, Not Adequately Controlled With Oral Vitamin D Receptor Activator (Calcitriol or Alfacalcidol)
Brief Title: Study of Zemplar iv in Patients With End Stage Chronic Kidney Disease, Undergoing Haemodialysis
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: P10-231
Record Dates: First submitted 2010-02-22; First posted 2010-03-10 (Estimated); Results first posted 2011-09-12 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Parathyroid Hormone
Keywords: paricalcitol iv; vitamin D; secondary hyperparathyroidism; hemodialysis
MeSH Terms: conditions — Hyperparathyroidism, Secondary

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- End stage chronic kidney disease: Secondary hyperparathyroidism defined as intact PTH > 300 pg/mL
  Interventions: Drug: Zemplar iv (paricalcitol iv)

INTERVENTIONS:
Drug: Zemplar iv (paricalcitol iv) — Each patient will be treated at the physician's discretion. Zemplar (paricalcitol) will be prescribed in the usual manner in accordance with the approved Summary of Product Characteristics.
  Other Names: Zemplar iv

SUMMARY:
This is the post-marketing study conducted in two countries: Croatia and Serbia. In both countries Zemplar (paricalcitol) is the first injectable form of any Vitamin D Receptor (VDR) activator available for chronic kidney disease patients on hemodialysis. The evaluation of outcomes of VDR activator treatments in clinical practice is a major challenge in the management of this patient population. The aim of this post-marketing observational study is to obtain further data on the outcomes of Zemplar Injection administration during routine clinical use.

DETAILED DESCRIPTION:
This study is a non-interventional, observational study in which Zemplar® Injection is prescribed in the usual manner in accordance with the terms of the local Summary of Product Characteristics (SmPC) with regards to dose, population and indication. The study population consists of participants receiving hemodialysis in whom the diagnosis of secondary hyperparathyroidism has been established, and who are not adequately controlled with the oral VDR activator (calcitriol or alfacalcidol). Participants will be included via consecutive sampling. To be included, participants should have a clinical indication to initiate treatment with Zemplar® Injection due to: (1) a diagnosis of secondary hyperparathyroidism and (2) because they require a change in treatment for secondary hyperparathyroidism (e.g. due to a lack of effectiveness of the previous treatment). Each participant will be observed during his/her Zemplar® Injection treatment regimen for a maximum period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject is more than 18 years of age and diagnosed with secondary hyperparathyroidism and has a pretreatment iPTH > 300 pg/mL, receiving chronic hemodialysis.
* Subject for which treatment with Zemplar Injection is indicated clinically according to the criteria of participating investigator.

Exclusion Criteria:

* Subject has a corrected serum calcium >10.5 mg/dL, serum phosphorus > 6.5 mg/dL or subjects with corrected Ca x P>65.
* Subject has known hypersensitivity and/or toxicity to vitamin D metabolites and/or other product ingredients, or has participated in clinical study within the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Haemodialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2007-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Gunjaca, MD, Study Director — Abbott
Locations (21):
- Croatia (14):
  - Site Reference ID/Investigator# 27525, Dubrovnik
  - Site Reference ID/Investigator# 27531, Imotski
  - Site Reference ID/Investigator# 6175, Karlovac
  - Site Reference ID/Investigator# 27528, Pula
  - Site Reference ID/Investigator# 27533, Rijeka
  - Site Reference ID/Investigator# 27523, Sisak
  - Site Reference ID/Investigator# 27529, Slavonski Brod
  - Site Reference ID/Investigator# 27530, Split
  - Site Reference ID/Investigator# 27524, Šibenik
  - Site Reference ID/Investigator# 27534, Trogir
  - Site Reference ID/Investigator# 27522, Vinkovci
  - Site Reference ID/Investigator# 27527, Zadar
  - Site Reference ID/Investigator# 27526, Zagreb
  - Site Reference ID/Investigator# 27532, Zagreb
- Serbia (7):
  - Site Reference ID/Investigator# 27536, Belgrade
  - Site Reference ID/Investigator# 27538, Belgrade
  - Site Reference ID/Investigator# 27539, Belgrade
  - Site Reference ID/Investigator# 6169, Belgrade
  - Site Reference ID/Investigator# 27540, Belgrade
  - Site Reference ID/Investigator# 27535, Bor
  - Site Reference ID/Investigator# 27537, Kragujevac

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Safety population consists of 181 participants who received at least one dose of drug. Of those, 175 were included in the full analysis set. Six participants were excluded; five due to initial intact parathyroid hormone values less than 300 picograms per milliliter and one suffered a serious adverse event before the first evaluation (study visit).
Groups:
- End Stage Chronic Kidney Disease: Participants receiving hemodialysis for end stage chronic kidney disease in whom a diagnosis of secondary hyperparathyroidism (defined as intact parathyroid hormone [iPTH] less than 300 picograms per milliliter [pg/mL]) has been established. Zemplar (paricalcitol) injection was to be prescribed in the usual manner in accordance with the terms of the local Summary of Product Characteristics.
Period: Overall Study
Arm/Group | End Stage Chronic Kidney Disease
Started | 181
Completed | 113
Not Completed | 68
Not completed — Drug not available | 30
Not completed — Adverse Event | 9
Not completed — Kidney transplant | 6
Not completed — Serious Adverse Event | 3
Not completed — Lack of effectiveness | 2
Not completed — Patient noncompliance | 2
Not completed — Hyperphosphatemia | 2
Not completed — Nodular hyperplasia of parathyroid gland | 2
Not completed — Change of residence | 2
Not completed — Over-suppression of parathyroid gland | 2
Not completed — Reason unknown | 8

BASELINE CHARACTERISTICS:
Arm/Group | End Stage Chronic Kidney Disease
Number analyzed (Participants) | 175
Age Continuous [Mean (Standard Deviation); unit: years] | 55.3 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 96

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving at Least a 40% Reduction of iPTH (Intact Parathyroid Hormone) From Baseline
Time Frame: Baseline through 12 months
Population: Of the 175 participants in the full analysis set, one participant was excluded from the analysis due to missing data.
Measure: Number; unit: percentage of participants
Arm/Group | End Stage Chronic Kidney Disease
Number analyzed (Participants) | 174
percentage of participants | 58.1

2. Secondary Outcome: Percentage of Subjects Achieving Serum iPTH Level Less Than or Equal to 300 Picograms Per Milliliter (pg/mL)
Description: Percentage of subjects achieving a serum iPTH level less than or equal to 300 pg/mL on the final visit.
Time Frame: Baseline through 12 months
Population: Of the 175 participants in the full analysis set, one participant was excluded from the analysis due to missing data.
Measure: Number; unit: percentage of participants
Arm/Group | End Stage Chronic Kidney Disease
Number analyzed (Participants) | 174
percentage of participants | 43.7

3. Secondary Outcome: Time (Measured in Days) to Achieve Intact Parathyroid Hormone (iPTH) Levels Less Than or Equal to 300 pg/mL
Description: The average time (measured in days) to achieve target iPTH levels.
Time Frame: Baseline through 12 months
Population: Of the 175 participants in the full analysis set, one participant was excluded from the analysis due to missing data.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | End Stage Chronic Kidney Disease
Number analyzed (Participants) | 174
Days | 107.0 (102.7)

4. Secondary Outcome: Clinically Meaningful Hypercalcemia, Defined as Corrected Serum Calcium Greater Than 11.0 Milligrams Per deciLiter (mg/dL) Taken at Two Consecutive Measurements.
Description: Number of participants with clinically meaningful hypercalcemia, defined as corrected serum calcium greater than 11.0 milligrams per deciLiter (mg/dL) taken at two consecutive measurements (visits) during the study.
Time Frame: Baseline through 12 months
Population: Analysis was based on the number of subjects included in the full analysis set (N=175).
Measure: Number; unit: participants
Arm/Group | End Stage Chronic Kidney Disease
Number analyzed (Participants) | 175
participants | 2

ADVERSE EVENTS:
Time Frame: Study start for up to 12 months (end of study). All serious adverse events were reported from the time the physician obtained the patient's authorization to use and disclose information (informed consent).
Description: Serious adverse events were assessed at each study visit. Adverse events with an onset date on or after the day of first dose and up to 30 days after the last dose of Zemplar (paricalcitol) therapy were summarized.
Arm/Group | End Stage Chronic Kidney Disease
Serious Adverse Events (participants affected / at risk) | 15/181
Other Adverse Events (participants affected / at risk) | 20/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | End Stage Chronic Kidney Disease (N=181)
Cardiopulmonary arrest (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 2
Pulmonary edema (Cardiac disorders) | 1
Parathyroid adenoma (Endocrine disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Paresis (Nervous system disorders) | 1
Spinal cord neoplasm (Nervous system disorders) | 1
Death (General disorders) | 1 — Reason for death is unknown, assessed as not related to study drug.
Bronchopneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Cancer of lung (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Vascular disorders) | 1
Radial artery embolism (Vascular disorders) | 1
Thrombosis arteriovenous fistula (Vascular disorders) | 1
Gastritis chronic (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | End Stage Chronic Kidney Disease (N=181)
Hypercalcemia (Endocrine disorders) | 13
Hyperphosphaetemia (Endocrine disorders) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.